CLINICAL TRIAL: NCT03255499
Title: Efficacy of the MovinCog Intervention in Children: A Randomized, Placebo-controlled Trial
Brief Title: Efficacy of the MovinCog Intervention in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, David Moreau, PhD, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC081017
Record Dates: First submitted 2017-08-11; First posted 2017-08-21 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Learning Disorders; Learning Disabilities; Cognitive Change
Keywords: cognitive training; physical exercise; brain dynamics; cognitive abilities; physiological markers
MeSH Terms: conditions — Learning Disabilities; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise and cognitive training (Experimental): This intervention includes a combination of high-intensity exercise (10min/day) and computerized cognitive training (20min/day). The software for the latter has been developed by our group, and includes 8 mini-games targeting different cognitive abilities. Both are developed for the MovinCog intervention. The intervention is personalized, based on individual performance.
  Interventions: Behavioral: Exercise; Behavioral: Cognitive
- Exercise (Experimental): High-intensity training regimen, 10min/day. Developed for the MovinCog intervention.
  Interventions: Behavioral: Exercise
- Cognitive training (Experimental): Computerized cognitive training, 20min/day. Developed for the MovinCog intervention.
  Interventions: Behavioral: Cognitive
- Games (Active Comparator): The active control is composed of a blend of board games, computer games, and trivia quizzes. Specific content is personalized based on individual preferences, so as to reflect the flexibility of the experimental arms.
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Exercise — Exercise
  Arms: Exercise; Exercise and cognitive training
Behavioral: Cognitive — Cognitive
  Arms: Cognitive training; Exercise and cognitive training
Behavioral: Active control — Active control, including a blend of computer games, board games, quizzes, trivia
  Arms: Games

SUMMARY:
This study aims to test the efficacy of the MovinCog Intervention to enhance cognitive abilities in children 7-15 yrs. The intervention consists of two parts: a physical exercise regimen, based on high-intensity training, and a cognitive training component. The design will contrast the intervention with an active control group, matched for expectancy effects.

DETAILED DESCRIPTION:
Specifically, the investigators will compare both components together (exercise and cognitive training) against either one of the components (exercise alone, or cognitive training alone) and against an active control group. The study will include measures of scholastic aptitude, as well as of working memory and cognitive control (primary outcome measures), two cognitive abilities that are critical to daily life activities, and that respond well to training. In addition, the investigators will measure physiological responses to training, to monitor changes associated with exercise (secondary outcome measures). Finally, the investigators will relate training-specific improvements with transfer gains, to better model the interaction between training and transfer. This will provide a comprehensive understanding of the dynamics associated with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-15

Exclusion Criteria:

* Age outside inclusion criteria
* History of seizures, brain trauma

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2017-09-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline working memory capacity at 10 weeks | Baseline and 10-week posttest
  Constructs measured by multiple tasks (bds, corsi, n-back)
Change from baseline cognitive control at 10 weeks | Baseline and 10-week posttest
  Constructs measured by multiple tasks (flanker, go/no-go, stroop)
Change from baseline scholastic aptitude at 10 weeks | Baseline and 10-week posttest
  Constructs measured by multiple national (New Zealand), standardized tests

SECONDARY OUTCOMES:
Change from baseline resting heart rate at 10 weeks | Baseline and 10-week posttest
  Measured by monitor
BDNF polymorphism measured by genetic saliva kit | Baseline
  Effect of BDNF polymorphism on primary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: David Moreau, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Release IPD at the time of publication.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Post-publication
Access Criteria: Unrestricted
URL: http://github.com/davidmoreau/

REFERENCES:
- [Derived] Moreau D, Kirk IJ, Waldie KE. High-intensity training enhances executive function in children in a randomized, placebo-controlled trial. Elife. 2017 Aug 22;6:e25062. doi: 10.7554/eLife.25062. PMID 28825973